CLINICAL TRIAL: NCT03742271
Title: Evaluation of Senofilcon A With New UV-blocker on a Neophyte Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-6241
Record Dates: First submitted 2018-11-13; First posted 2018-11-15 (Actual); Results first posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-02

CONDITIONS: Visual Acuity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- senofilcon A (Experimental): Subjects that are habitual spectacle wearers that have never worn contact lenses and have had an eye exam and an updated spectacle prescription in the last 6 months will be enrolled and fitted into the senofilcon A TEST Lens for a total period of 4 weeks.
  Interventions: Device: senofilcon A

INTERVENTIONS:
Device: senofilcon A — TEST Lens

SUMMARY:
This is a 5-visit, single-arm, open-label, dispensing study. Each subject will be bilaterally fit with the test article for approximately 4 weeks of reusable daily wear with lens replacement occurring 2-weeks after initial dispensing. After 4 weeks of study lens wear, subjects will return to their habitual spectacles for one week.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

  1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. Between 18 and 39 (inclusive) years of age at the time of screening.
  4. They are a contact lens 'neophyte'. In this work 'neophyte' is taken to mean any subject who has never been dispensed contact lenses. A subject who had taken part in a non-dispensing clinical study or had been fitted with contact lenses in practice but never went on to actually wear the lenses, is also classified as a 'neophyte'.
  5. Habitual spectacles must have resulted from an eye exam within the past six months.
  6. The subject must have worn the updated spectacles for at least two weeks.
  7. Be a current wearer of prescription spectacles that provide corrected monocular visual acuity of 20/25 or better in each eye.
  8. The subject's vertex corrected spherical equivalent distance refraction must be in the range of -1.00 to -6.00 D (inclusive) in each eye.
  9. The subject's refractive cylinder must be -1.00 D or less in each eye.
  10. Have spherocylindrical best corrected distance Snellen visual acuity of 20/25 or better in each eye.

      Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating

  1. Currently pregnant or lactating.
  2. Any active or ongoing systemic disease (e.g., Sjögren's Syndrome), allergies, infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive diseases (e.g., HIV), autoimmune disease (e.g. rheumatoid arthritis), or other diseases, by self-report, which are known to interfere with contact lens wear and/or participation in the study.
  3. Use of systemic medications that have a high likelihood to interfere with contact lens wear (estrogens, antihistamines, anticholinergics, beta-blockers, and psychotropics).
  4. Any current use of ocular medication.
  5. Any known hypersensitivity or allergic reaction to any ingredient in Opti-Free PureMoist.
  6. Any previous or planned (during the course of the study) ocular surgery (e.g., radial keratotomy, PRK, LASIK, etc.).
  7. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
  8. Any ocular allergies, infections or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or corneal distortion.
  9. Any Grade 3 or 4 slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA slit lamp classification scale.
  10. Binocular vision abnormality or strabismus.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Vue Optical Boutique, Jacksonville, Florida
  - Atlantic Eye Institute, Jacksonville Beach, Florida
  - Sabal Eye Care, Longwood, Florida
  - Baker Vision Care, Macclenny, Florida
  - Georgia Center for Sight, Greensboro, Georgia
  - Advanced Eyecare, Raytown, Missouri
  - ABQ Eye Care, Albuquerque, New Mexico
  - Sacco Eye Group, Vestal, New York
  - ProCare Vision Centers, Granville, Ohio
  - Eyecare Professionals of Powell, Powell, Ohio
  - Frazier Vision Inc., Tyler, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 129 subjects were enrolled in this study. Of those enrolled, 127 subjects were assigned and dispensed the Test lens while, 2 subjects failed to meet all eligibility criteria. Of those dispensed, 115 subjects completed the study while, 12 subjects were discontinued from the study.
Groups:
- Senofilcon A: All subjects wore the senofilcon A lens for the first 4-Weeks of the study and then wore their Habitual spectacles for a period of 1-Week after the 4-Weeks of lens wear.
Period: Overall Study
Arm/Group | Senofilcon A
Started | 127
Completed | 115
Not Completed | 12
Not completed — Unsatisfactory Visual Response | 1
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 4
Not completed — Failed Insertion & removal | 3
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Groups:
- All Dispensed Subjects: All subjects dispensed the senofilcon A lens during any point in the study.
Arm/Group | All Dispensed Subjects
Number analyzed (Participants) | 127
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.3 (5.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71
  Male | 56
Race/Ethnicity, Customized [Number; unit: Count of Participants]
  Asian | 4
  American Indian or Alaska Native | 1
  Black or African American | 16
  White | 101
  Other | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 127

OUTCOME MEASURES:

1. Primary Outcome: Acceptable Lens Fitting
Description: Acceptable fit is determined by the eye care practitioner (ECP/investigator) and includes the following criteria; (1) physiological responses (No Grade 3 or higher slit lamp findings), (2) mechanical lens fitting (no unacceptable lens fitting in either eye), (3) subjects' assessment of comfort, vision and handling.
Time Frame: 4-Week Follow-up
Population: All subjects who were administered a Test lens and completed through the 4-week evaluation in which the eye care practitioner completed the lens fitting assessment.
Measure: Number; unit: Proportion of subjects
Groups:
- Senofilcon A: All subjects in this study wore the senofilcon A lens in both eyes through the 4-Week follow-up evaluation
Arm/Group | Senofilcon A
Number analyzed (Participants) | 114
Proportion of subjects | 0.974
Statistical Analysis 1: Comparison: Senofilcon A; This study was powered to test the hypothesis that at least 50% will have an acceptable lens fitting; Test type: Superiority — Superiority was concluded in the lower limit of the 95% confidence interval was above 0.50; Binomial Exact Test; Proportion = 0.974, 95% CI 2-sided [0.925 to 0.995]

ADVERSE EVENTS:
Time Frame: Approximately 4 weeks per subject.
Groups:
- Senofilcon A: All subjects that wore the senofilcon A lens in either eye during any point of the study.
Arm/Group | Senofilcon A
All-Cause Mortality (participants affected / at risk) | 0/127
Serious Adverse Events (participants affected / at risk) | 0/127
Other Adverse Events (participants affected / at risk) | 0/127

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-10-11): https://cdn.clinicaltrials.gov/large-docs/71/NCT03742271/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-13): https://cdn.clinicaltrials.gov/large-docs/71/NCT03742271/SAP_001.pdf